CLINICAL TRIAL: NCT02480907
Title: Supporting Carers of Children and Adolescents With Eating Disorders in Austria (SUCCEAT) - A Randomized Controlled Trial to Compare Workshop, Internet-based and Conventional Parental Support Groups
Brief Title: Supporting Carers of Children and Adolescents With Eating Disorders in Austria (SUCCEAT)
Acronym: SUCCEAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Pharmig - Gesundheitsziele aus dem Rahmen-Pharmavertrag (Other)
Responsible Party: Principal Investigator, Dr. Andreas Karwautz, Univ. Prof. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FA765A0304
Record Dates: First submitted 2015-04-07; First posted 2015-06-25 (Estimated); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Mental Health
Keywords: eating disorders; caregivers; parents; skills training; workshops; support; internet; online; family
MeSH Terms: conditions — Psychological Well-Being; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Workshop Group (Active Comparator): Parents of ~ 40 children and adolescents within the age group of 10-18 years suffering from anorexia or bulimia nervosa will be involved in the workshop support group for parents for a period of three months, including a written manual, a DVD (Digital Video Disc) with additional information and weekly workshops. Over the course of three months, parents will participate at the 8 workshop sessions and get the manual to read and the DVDs to use at home to illustrate workshop contents with examples and video clips.
  Interventions: Behavioral: Workshop Group
- Internet-based support group (Active Comparator): Parents of ~ 40 children and adolescents within the age group of 10-18 years suffering from anorexia or bulimia nervosa will be involved in the Internet-based support group for parents, including material from the manual and the DVD and additional information available online within a structured program. Over the course of three months, parents will get access to the 8 support sessions online with the instruction to work out the program at home. Additionally email support is offered after completing each session.
  Interventions: Behavioral: Internet-based support group
- Control group - TAU (No Intervention): Parents of ~ 40 children and adolescents within the age group of 10-18 years suffering from anorexia or bulimia nervosa will get treatment as usual and take part in conventional parental intervention groups.

INTERVENTIONS:
Behavioral: Workshop Group — Workshop support group
  Arms: Workshop Group
Behavioral: Internet-based support group — Internet based support group with E-mail coaching
  Arms: Internet-based support group

SUMMARY:
The purpose of the "Supporting Carers of Children and Adolescents with Eating Disorders in Austria" (SUCCEAT) - study is to compare Workshop, Internet-based and Conventional Parental Support Groups for carers of chilren and adolescents between 10 and 18 years in a randomized controlled trial for the first time in Austria.

DETAILED DESCRIPTION:
According to NICE guidelines, eating disordered patients should be managed on an outpatient basis. This challenge seems to put a heavy burden on most caregivers. Schmidt and Treasure (2006) argued that obsessive compulsive personality traits, emotional avoidance, pro-anorectic beliefs and responses of close others like dysfunctional communication styles impair the outcome. The construct of expressed emotions reflects on the amount of criticism, hostility and emotional over-involvement expressed by relatives of psychiatric patients towards them. A special program for parents is developed to equip caregivers with knowledge and skills to change maintaining factors and therefore improve the patient's outcome. Furthermore coping strategies are provided to help carers to reduce their burden. We start a randomized controlled trial comparing two interventions with a conventional group. We compare Workshops (Intervention Group 1), Internet-based (Intervention Group 2) and Conventional (Control Group) Carers´ Support Groups. Before starting the intervention (T0, baseline), at the end of the intervention (T1) and 1 year after the intervention (T2, follow up) assessments will be conducted via questionnaires and interviews. Parents of 48 children and adolescents within the age group of 10-17 years suffering from anorexia or bulimia nervosa will be involved in each group, resulting in an overall sample size of 144. The investigators aim is to equip parents with knowledge and skills in order to support their children's recovery, prevent relapse and improve their own wellbeing. The long term goal is to provide low-threshold, cost-effective, time-efficient and superregional support for parents in the future.

ELIGIBILITY:
Inclusion Criteria:

* children and adolescents aged 10-18, who suffer from anorexia or bulimia nervosa and their primary caregivers

Exclusion Criteria:

* no written informed consent possible due to intelligence or no willingness by parents to include minor

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 144 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2019-03-05 (Actual); Study Completion 2019-03-05 (Actual)

PRIMARY OUTCOMES:
Psychological morbidity and distress in caregivers are measured with the "Gerneral Health Questionnaire - 12" | 15 months
  Questionnaire

SECONDARY OUTCOMES:
Emotional problems in caregivers will be measured with the "Beck Depression Inventory" (measures the severity of Depression) | 15 months
  Questionnaire
Emotional problems in caregivers will be measured with the "State- Trait Anxiety Inventory" | 15 months
  Questionnaire
Emotional Problems will be measured with the "The Family-Questionnaire" (measures the emotional climate within the Family) | 15 months
  Questionnaire
Emotional problems in caregivers will be measured with the "Symptom Checklist-90-Revised" (measures psychological problems and symptoms of psychopathology) | 15 months
  Questionnaire
Behavioral and social problems in caregivers will be measured with the "Caregiver Skills Scale" (measures caregiver skills that may be helpful in supporting people with anorexia nervosa) | 15 months
  Questionnaire
Behavioral and social problems in caregivers will be measured with the "Eating Disorder Symptom Impact Scale" (measures which impact the eating disorder symptoms of the patient have upon the well-being of the caregiver) | 15 months
  Questionnaire
Behavioral and social problems in caregivers will be measured with the german Version of the "University of Rhode Island Change Assessment Scale " (= Fragebogen zur Erfassung der Veränderungsbereitschaft) (measures stages of Change) | 15 months
  Questionnaire
Needs of carers will be measured with the "Carers' Needs Assessment Measure" (measures the needs of carers of patients with an eating disorder) | 15 months
  Questionnaire
Caregiving appraisal will be measured with the "Experience of Caregiving Inventory" (measures general aspects of care giving experiences) | 15 months
  Questionnaire
Behavioural and emotional problems in patients are measured via the "Youth self Report" | 15 months
  Questionnaire
Emotional Problems in patients are measured via the "Family Emotional Involvement and Criticism Scale" (measures expressed emotions) | 15 months
  Questionnaire
Emotional Problems in patients are measured via the german questionnaire "Fragebogen zur gesundheitsbezogenen Lebensqualität bei Kinder und Jugendlichen" (measures life-Quality; only available in german). | 15 months
  Questionnaire
The presence of the eating disorder in the patients will be measured via the "Eating Disorder Examination" (measures the range and severity of the eating disorder components) | 15 months
  Interview
The presence of the eating disorder in the patients will be measured via the "Anorexia Nervosa/Bulimia Nervosa Stages of Change Questionnaire" (measures the motivation to change in the patients with an eating disorder) | 15 months
  Questionnaire
Feasibility and Acceptability of the workshops and online modules (Treatment Satisfaction Questionnaire, developed by our research group) | 15 months
  Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Karwautz, MD, Prof, Study Director — Medical University Vienna; Gudrun Wagner, Mag, Dr, Study Director — Medical University Vienna
Locations (1):
- Medical University of Vienna, Dep. of Child and Adolescent Psychiatry, Vienna, Austria

REFERENCES:
- [Derived] Franta C, Philipp J, Waldherr K, Truttmann S, Merl E, Schofbeck G, Koubek D, Laczkovics C, Imgart H, Zanko A, Zeiler M, Treasure J, Karwautz A, Wagner G. Supporting Carers of Children and Adolescents with Eating Disorders in Austria (SUCCEAT): Study protocol for a randomised controlled trial. Eur Eat Disord Rev. 2018 Sep;26(5):447-461. doi: 10.1002/erv.2600. Epub 2018 May 6. PMID 29732651
- See also: related Information — http://www.ess-stoerung.eu